CLINICAL TRIAL: NCT06523816
Title: Correlation Between Dermoscopy and Histopathology in Non-melanocytic Skin Tumors
Brief Title: Dermoscopy and Histopathology in Non-melanocytic Skin Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaza Alaa Ezzat Abdel-moneim, Resident, Assiut University
Other Study IDs: NMSTs
Record Dates: First submitted 2024-07-23; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Non-melanoma Skin Cancer
MeSH Terms: interventions — Dermoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: dermoscopy — Dermoscopy is a fast imaging technique that allows an excellent visualization of non-melanocytic skin tumors to diagnose them without invasive interventon.

SUMMARY:
The main aim of the study is to investigate the relation between dermoscopic findings in pre-operative diagnosis of non-melanocytic skin tumors and post-operative histopathology findings .

ELIGIBILITY:
Inclusion Criteria:

* All patients with NMST clinically of both genders in all ages with positive dermoscopic findings and definite histopathologic diagnosis of NMST

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from those attending the outpatient clinic of department of Dermatology , Assiut University Hospitals.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity of dermoscopy to detect NMSTs | 2 years
  investigate the relation between dermoscopic findings in pre-operative diagnosis of non-melanocytic skin tumors and post-operative histopathology findings